CLINICAL TRIAL: NCT02128919
Title: Transcranial Direct Current Stimulation (tDCS) As A Treatment For Cigarette Craving and Cognitive Deficits in Schizophrenic
Acronym: TDCSSCHIZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Robert C. Smith MD PhD, Research Psychiatrist, Nathan Kline Institute for Psychiatric Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 309320
Record Dates: First submitted 2014-04-26; First posted 2014-05-01 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia; Cognition; Cigarette Smoking
Keywords: Schizophrenia; Cigarette smoking; Cognition; Craving; MATRICS
MeSH Terms: conditions — Schizophrenia; Cigarette Smoking | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): tDCS 2 ma for 20 minutes with anode at DLPFC once a day for 5 days
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): tDCS 2 ma for 40 seconds with anode at DLPFC for 5 days
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Transcranial Direct Current Stimulation

SUMMARY:
This is a study of the effects of tDCS on smoking, craving for cigarettes, cognition, and psychiatric symptoms in schizophrenic patients who are current smokers or have a history of regular cigarette smoking. It assesses smoking with CO monitoring, nicotine and nicotine levels, and craving with QSU scale and response to craving slides. Cognition is measured by MCCB, symptoms are measured by PANSS and hallucination scale.

This is a double-blind sham-controlled study with active tDCS 2ma or 20 minutes over 5 days, and sham tDCS for 40 seconds on each sham occasion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia spectrum disorder History of cigarette smoking

Exclusion Criteria:

* Seizure disorder or current treated neurological illness Current Acute exacerbation of psychotic state

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Smith, MD, Principal Investigator — Nathsan Kline Institute for Psychiatric Research
Locations (1):
- Nathan Kline Institute for Psychiatric Research, Orangeburg, New York, United States

REFERENCES:
- [Result] Smith RC, Boules S, Mattiuz S, Youssef M, Tobe RH, Sershen H, Lajtha A, Nolan K, Amiaz R, Davis JM. Effects of transcranial direct current stimulation (tDCS) on cognition, symptoms, and smoking in schizophrenia: A randomized controlled study. Schizophr Res. 2015 Oct;168(1-2):260-6. doi: 10.1016/j.schres.2015.06.011. Epub 2015 Jul 17. PMID 26190299

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS: tDCS 2ma for 20 min with anode at DLPFC once a day for 5 days
  tDCS: Transcranial Direct Current Stimulation
- Sham tDCS: tDCS 2 ma for 40 second s with anode at DLPFC for 5 days
  tDCS: Transcranial Direct Current Stimulation
Period: Overall Study
Arm/Group | Active tDCS | Sham tDCS
Started | 17 | 16
Completed | 14 | 15
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS | Sham tDCS | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (11.1) | 44.9 (9.2) | 45.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 14 | 10 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race/ethnicity: white | 6 | 4 | 10
  race/ethnicity: black-African american | 10 | 9 | 19
  race/ethnicity: hispanic | 0 | 1 | 1
  race/ethnicity: other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cigarette Craving
Description: The Brief Questionnaire on Smoking Urges (QSU-Brief) was used to measure cigarette cravings. Scores ranged from a minimum of 1 ("Strongly Disagree") to a maximum of 7 ("Strongly Agree") and were determined by self-reported responses to 10 statements about having cravings for smoking. Scores closer to 1 after treatment would indicate a better outcome. Responses to each of the 10 items in the scale were summed for one total score. With 10 items on this scale with a range of scores from 1 to 7, on each occasion of rating the minimum score would be 7 and the maximum score would be 70.
Time Frame: Baseline and after 5 tDCs sessions (mean time 8.7[SD 2.7] days after basleine)
Population: Findings are based on31 subjects (15 active tDCS and 16 sham tDCS) who completed this QSU-Brief questionnaire in at baseline and after 5 tDCS sessions.. Complete sample who entered study and were randomized were 33 subjects 24 male and 9 female, but all subjects did not complete QSU brief rating scale..
Measure: Least Squares Mean (Standard Error); unit: Units on QSU-Brief Scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 16
Units on QSU-Brief Scale | 14.40 (3.57) | 11.00 (3.45)

2. Secondary Outcome: Change From Baseline in Cognitive Performance
Description: The MATRICS Consensus Cognitive Battery (MCCB) was used to measure cognitive performance. Seven Domain scores and a Composite score are calculated by the proprietary MCCB Computer Scoring Program from raw scores on 10 individually administered subtests. We used the revised MCCB program (beta version) which allows for calculation of Domain and Composite scores with missing data. The Domain T-scores are percentile-ranked and range from <20 (<0.1 percentile) to >80 (>99.9 percentile). The Composite scores are also percentile-ranked and range from <213 (T<20, <0.1 percentile) to >487 (T>80, >99.9 percentile). Higher scores after baseline represent better outcomes. Here we report difference scores from post-treatment and baseline with positive difference scores representing better outcomes.
Time Frame: Baseline and 1-3 days (mean 1.8 [SD 1.4] days after 5 tDCS sessions( mean 8.7 days after baseline)
Measure: Least Squares Mean (Standard Deviation); unit: MATRICS domain difference scores
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 14 | 16
MATRICS domain difference scores
  MATRICS Composite Diff Score | 3.47 (4.09) | -0.85 (4.08)
  MATRICS Working Memory Diff Score | 4.04 (5.70) | -3.29 (5.68)
  MATRICS Attention/Vigilance Diff Score | 4.25 (7.17) | -1.91 (7.17)

3. Other Pre Specified Outcome: Change From Baseline in Psychiatric Symptoms
Description: The Positive and Negative Syndrome Scale (PANSS) was used to measure psychiatric symptoms. Item scores ranged from 1 (Absent) to 6 (Severe) for symptoms on the Positive Scale (total subscale range: 7-42), the Negative Scale (total subscale range: 7-42), and the General Psychopathology Scale (total subscale range:16-96). All three subscales were summed for the PANSS total score (total scale range: 30-180). Scores closer to 30 after baseline represented better outcomes. Here we report difference scores from post-treatment and baseline with negative difference scores representing better outcomes.
Time Frame: Baseline and after 5 tDCS sessions
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Active tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 15
Units on a scale
  PANSS total diff score | -1.51 (8.01) | -2.37 (8.01)
  PANSS postive diff score | -1.70 (3.10) | -1.63 (3.10)
  PANSS Negative diff score | 1.06 (4.38) | 0.68 (4.38)

ADVERSE EVENTS:
Time Frame: fuyll course of study over 2 years
Arm/Group | Active tDCS | Sham tDCS
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No